CLINICAL TRIAL: NCT03631992
Title: Downshifting Sweet Preference and Added Sugar Intake During Snacking
Brief Title: Snacks, Smiles and Taste Preferences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Monell Chemical Senses Center (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 24653; R01DC016616 (NIH)
Record Dates: First submitted 2018-05-29; First posted 2018-08-15 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2023-12

CONDITIONS: Development, Child
Keywords: Children; Sugar; Taste; Snacking; Biomarker; Mothers

STUDY DESIGN:
Intervention Model Description: The intervention group will receive snacks lower in added sugar and sweetness (children) and educational lessons on dental care, food labels, added sugar, and portion size (mothers) whereas the control group will receive typical snacks (children) and educational lessons on portion size, sleep, screen time, and physical activity (mothers). Control group will receive the educational lessons of the intervention group at the end of the trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and outcome assessors will be blind to hypotheses and group assignment. Investigators will be blind to the group assignment during statistical analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Sweet (Experimental): Children in intervention group will be provided with daily snacks lower in added sugar and sweetness and their mothers will receive educational lessons on dental care, reading food labels, and nutrition that support the goals of reducing "sweet" exposure and added sugar intake.
  Interventions: Behavioral: Low Sweet
- Regular Sweet (Sham Comparator): Children in the regular sweet control group will be provided with common snacks fed to children of this age and mothers will be given education lessons on portion size, physical activity, sleep, screen time and, at the end of the trial, dental care.
  Interventions: Behavioral: Regular Sweet

INTERVENTIONS:
Behavioral: Low Sweet — Children in the experimental group get repeated exposure to lower sweet snacks and mothers get education lessons on dental care, reading food labels, portion size, and nutrition.
  Arms: Low Sweet
Behavioral: Regular Sweet — Children in sham comparator get typical snacks and mothers get education lessons on portion size, physical activity, sleep, and screen time.
  Arms: Regular Sweet

SUMMARY:
The research study is designed is to determine whether children's acceptance of low sugar snacks, most preferred level of sweet and salty taste, and dietary intake of added sugars changes after repeated exposure to snacks lower in sweetness when compared to the control group.

DETAILED DESCRIPTION:
This is a longitudinal, randomized, within- and between- subject study of children and their mothers to determine whether children's repeated exposure to snacks lower in sweetness and mothers' educational lessons about dental health and nutrition (intervention group) affects children's acceptance of low sugar snacks, most preferred level of sweet and salty taste, and dietary intake of added sugars when compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* English speaking mother 18 years or older
* Mother has primary responsibility for the eligible child's care
* Mother has primary responsibility for feeding the eligible child
* Mother is responsible for purchasing food for the family
* Mother must be willing to refrain from eating food and beverages high in added sugars in the eligible child's presence for the duration of the study

Exclusion Criteria:

* Child is in full-day daycare or school
* Child is currently on a special diet (e.g. weight management programs)
* Child has severe food allergies (e.g. gluten, peanuts)
* Child has medical conditions know to affect growth or eating (e.g. diabetes, cystic fibrosis)
* Mother is a current smoker

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Change is being assessed in the children's liking of snacks low in sweetness | From timepoint 0 (baseline Temple visit at start of intervention) to T1 (1 month), T2 (2 month), T3 (3 month), T4 (4 month, end of intervention) and T5 (5 month, which is 1 month post-intervention delay)
  Children's grouping of the taste of novel snacks as liked, ok, or disliked as determined by lab-based measurements of liking using a picture-based 3-point hedonic scale depicting "yummy", "yucky", and "just-okay" responses; following the grouping of snacks into these categories, snacks will be ranked for most liked to most disliked [range: 4-6].
Change is being assessed in the children's intake of snacks low in sweetness | From timepoint 0 (baseline Temple visit at start of intervention) to T1 (1 month), T2 (2 month), T3 (3 month), T4 (4 month= end of intervention) and T5 (5 month which is 1 month, post-intervention delay)
  Children's intake of novel snacks in grams using weighed intake methods and behavioral parameters of intake from digital recordings; higher intake and consummatory responses indicate greater acceptance.
Change is being assessed in dietary intake of energy from added sugar | From timepoint 0 (baseline Temple visit at start of intervention) to T1 (1 month), T2 (2 month), T3 (3 month), T4 (4 month, end of intervention) and T5 (5 month, which is 1 month post-intervention delay)
  Dietary intake (kcal/d) will be determined from Automated Self-Administered Recall System (ASA24) completed by mothers for her child and herself.

SECONDARY OUTCOMES:
Change is being assessed in levels of hair biomarker for added sugar intake | From timepoint 0 (baseline Temple visit at start of intervention) to T4 (4 month visit=end of intervention)
  Estimates of added sugar intake will be determined via stable isotope ratio mass spectrometry methods on hair samples collected at the start (T0) and end of 4-month intervention (T4)
Change is being assessed in liking-based dietary intake survey | From timepoint 0 (baseline Temple visit at start of intervention) to T1 (1 month), T2 (2 month), T3 (3 month), T4 (4 month, end of intervention) and T5 (5 month, which is 1 month post-intervention delay)
  Dietary intake of foods as determined by measurements of the degree of dislike or like for a variety of foods and beverages (e.g., sweet/fat, fruit, vegetables) as well as experiences and activities; range: -100 (maximal dislike) to 100 (maximal like)]. The items in a given category (e.g., fruits; sweets/fats; healthy foods) are combined and averaged [range: -100 to 100; higher numbers reflect greater liking and intake]. The preschool adapted liking survey (PALS) is used for children and the adult liking survey (ALS) is used for mothers
Monitoring of individual differences in parenting feeding styles | From timepoint 0 (baseline visit at start of intervention) to T1 (1 month), T2 (2 month), T3 (3 month), T4 (4 month, end of intervention) and T5 (5 month, which is 1 month post-intervention delay)
  Mothers will complete the 19-item Child Feeding Styles and Practices Questionnaire [CFSQ]. Each item is scored from 1 (never) to 5 (always). Scores are averaged and categorized into one of four feeding styles: authoritative, authoritarian, indulgent and uninvolved; higher scores represent more of the feeding style
Monitoring of individual differences in children's appetitive drive | From timepoint 0 (baseline visit at start of intervention) to T1 (1 month), T2 (2 month), T3 (3 month), T4 (4 month, end of intervention) and T5 (5 month, which is 1 month post-intervention delay)
  Mothers will complete the 26-item Children's Eating Behavior Questionnaire [CEBQ]. Each item is scored from 1 (never) to 5 (always) and are averaged and categorized into aspects of child eating (e.g., enjoyment of food, food responsiveness, satiety responsiveness, emotional overeating; emotional undereating, food fussiness); higher numbers reflect more of the behavior
Monitoring of individual differences in children's palatable eating motivation | From timepoint 0 (baseline visit at start of intervention) to T1 (1 month), T2 (2 month), T3 (3 month), T4 (4 month, end of intervention) and T5 (5 month, which is 1 month post-intervention delay)
  Mothers will complete the 19-item Kids Palatable Eating Motive Scales (KPEMS) questionnaire; each item is scored from 1 (child almost never/never exhibits behavior) to 5 (child almost always/always exhibits behavior). Scores are averaged and categorized to reflect motives for intake of palatable foods (e.g., to socialize, cope, fit in or conform, for reward enhancement); higher numbers reflect more of the motivation
Monitoring of individual differences in mothers' palatable eating motivation | From timepoint 0 (baseline visit at start of intervention) to T1 (1 month), T2 (2 month), T3 (3 month), T4 (4 month, end of intervention) and T5 (5 month, which is 1 month post-intervention delay)
  Mothers will complete the 19-item Palatable Eating Motive Scales (PEMS) questionnaire; each item is scored from 1 (almost never/never exhibits behavior) to 5 (almost always/always exhibits behavior). Scores are averaged and categorized to reflect motives for intake of palatable foods (e.g., to socialize, cope, fit in or conform, for reward enhancement); higher numbers reflect more of the motivation
Monitoring of weight | From timepoint 0 (baseline visit at start of intervention) to T1 (1 month), T2 (2 month), T3 (3 month), T4 (4 month= end of intervention) and T5 (5 month which is 1 month, post-intervention delay)
  Children's weight will be measured in kg; these measures will be converted to weight for age Z scores which provide measures of anthropometry adjusted age and sex.
Monitoring of height | From timepoint 0 (baseline visit at start of intervention) to T1 (1 month), T2 (2 month), T3 (3 month), T4 (4 month= end of intervention) and T5 (5 month which is 1 month, post-intervention delay)
  Children's height will be measured in cm; these measures will be converted to height for age Z scores which provide measures of anthropometry adjusted age and sex.
Monitoring of body mass index | From timepoint 0 (baseline visit at start of intervention) to T1 (1 month), T2 (2 month), T3 (3 month), T4 (4 month= end of intervention) and T5 (5 month which is 1 month, post-intervention delay)
  Children's height will be measured in cm and weight in kg; these measures will be combined to determine BMI (kg/m2) and then converted to BMI Z scores which provide measures of anthropometry adjusted age and sex.

OTHER OUTCOMES:
Concordance of hair biomarker for added sugar intake among mother-child dyads | Relationship between hair biomarker levels at timepoint 0 (baseline Temple visit at start of intervention) and at T4 (4 month visit=end of intervention)
  Estimates of added sugar intake will be determined via stable isotope ratio mass spectrometry methods on hair samples collected from mother and child at the start (T0) and end of 4-month intervention (T4) end of the 4-month intervention period (T4) to determine concordance among mother-child dyads

CONTACTS AND LOCATIONS:
Overall Officials: Julia Mennella, PhD, Principal Investigator — Monell Chemical Senses Center; Jennifer O Fisher, PhD, Principal Investigator — Temple University
Locations (2):
- United States (2):
  - Monell Chemical Senses Center, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
dbGAP
Supporting Information: Study Protocol, SAP
Time Frame: 2022 and for one year
Access Criteria: To be developed

REFERENCES:
- [Background] Mennella JA, Lukasewycz LD, Griffith JW, Beauchamp GK. Evaluation of the Monell forced-choice, paired-comparison tracking procedure for determining sweet taste preferences across the lifespan. Chem Senses. 2011 May;36(4):345-55. doi: 10.1093/chemse/bjq134. Epub 2011 Jan 12. PMID 21227904
- [Background] Nash SH, Kristal AR, Hopkins SE, Boyer BB, O'Brien DM. Stable isotope models of sugar intake using hair, red blood cells, and plasma, but not fasting plasma glucose, predict sugar intake in a Yup'ik study population. J Nutr. 2014 Jan;144(1):75-80. doi: 10.3945/jn.113.182113. Epub 2013 Nov 6. PMID 24198311
- [Background] Mennella JA, Finkbeiner S, Lipchock SV, Hwang LD, Reed DR. Preferences for salty and sweet tastes are elevated and related to each other during childhood. PLoS One. 2014 Mar 17;9(3):e92201. doi: 10.1371/journal.pone.0092201. eCollection 2014. PMID 24637844
- [Background] Wardle J, Guthrie CA, Sanderson S, Rapoport L. Development of the Children's Eating Behaviour Questionnaire. J Child Psychol Psychiatry. 2001 Oct;42(7):963-70. doi: 10.1111/1469-7610.00792. PMID 11693591
- [Background] Vandeweghe L, Verbeken S, Moens E, Vervoort L, Braet C. Strategies to improve the Willingness to Taste: The moderating role of children's Reward Sensitivity. Appetite. 2016 Aug 1;103:344-352. doi: 10.1016/j.appet.2016.04.017. Epub 2016 Apr 19. PMID 27103060
- [Background] Hughes SO, Power TG, Orlet Fisher J, Mueller S, Nicklas TA. Revisiting a neglected construct: parenting styles in a child-feeding context. Appetite. 2005 Feb;44(1):83-92. doi: 10.1016/j.appet.2004.08.007. Epub 2004 Nov 13. PMID 15604035
- [Background] Sharafi M, Rawal S, Fernandez ML, Huedo-Medina TB, Duffy VB. Taste phenotype associates with cardiovascular disease risk factors via diet quality in multivariate modeling. Physiol Behav. 2018 Oct 1;194:103-112. doi: 10.1016/j.physbeh.2018.05.005. Epub 2018 May 8. PMID 29746892
- [Background] Martignon S, Gonzalez MC, Tellez M, Guzman A, Quintero IK, Saenz V, Martinez M, Mora A, Espinosa LF, Castiblanco GA. Schoolchildren's tooth brushing characteristics and oral hygiene habits assessed with video-recorded sessions at school and a questionnaire. Acta Odontol Latinoam. 2012;25(2):163-70. PMID 23230636
- [Background] Mennella JA, Pepino MY, Lehmann-Castor SM, Yourshaw LM. Sweet preferences and analgesia during childhood: effects of family history of alcoholism and depression. Addiction. 2010 Apr;105(4):666-75. doi: 10.1111/j.1360-0443.2009.02865.x. Epub 2010 Feb 9. PMID 20148789
- [Derived] Smethers AD, Fisher JO, Carney EM, Coffman DL, Mennella JA. Carbon stable isotope values in hair are associated with added sugar intake in adults but not young children: a cross-sectional study. Am J Clin Nutr. 2025 Apr;121(4):900-909. doi: 10.1016/j.ajcnut.2025.02.013. Epub 2025 Feb 18. PMID 39978470